CLINICAL TRIAL: NCT05504915
Title: Prospective, Non-interventional, Observational Study in Cohort of Patients With IBD at University Hospital Center Osijek Switching From IV to SC Vedolizumab to Observe Vedolizumab Serum Concentration and Treatment Outcomes
Brief Title: Real World Data on Vedolizumab Concentration and Outcomes in Inflammatory Bowel Disease (IBD) Patients Switching From Intravenous (IV) to Subcutaneous (SC) Vedolizumab in University Hospital Center Osijek
Status: Completed | Type: Observational
Sponsor: Osijek University Hospital (Other)
Collaborators: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Vlasta Orsic Fric, Principal Investigator, Osijek University Hospital
Other Study IDs: DGH01
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with IBD: Participants diagnosed with IBD (UC or CD) who switched from vedolizumab IV to vedolizumab SC treatment during routine clinical practice, will be observed prospectively for up to 12 months from switch.

SUMMARY:
Inflammatory bowel disease consists of ulcerative colitis (UC) or Crohn's disease (CD). The main aim of this study is to describe real-world data on vedolizumab serum concentration and treatment outcomes in cohort of patients treated at the Department of Gastroenterology and Hepatology of University Hospital Center Osijek. Study will be recruiting patients who switched from intravenous to subcutaneous vedolizumab according to routine clinical practice.

DETAILED DESCRIPTION:
This is a non-interventional, prospective study of participants with IBD who switched from intravenous to subcutaneous vedolizumab in the real world setting.

The study will enroll approximately 30 participants. The data will be collected at the Department of Gastroenterology and Hepatology of University Hospital Center Osijek. All the participants will be assigned to a single observational cohort. All procedures (e.g., blood draw for serum trough concentration of vedolizumab, stool collection for fecal calprotectin or colonoscopy) will be done for routine clinical care. Data will be collected at baseline and at 6-12 months after switch from intravenous to subcutaneous vedolizumab. At baseline, data on age, gender, body mass, diagnosis, time from diagnosis, prior and concomitant therapy for IBD, comorbidities, time from switch from vedolizumab IV to vedolizumab SC, and vedolizumab serum trough concentration during vedolizumab IV therapy, will be collected. At control visit, data on concomitant therapy, adverse events, hospitalization, surgery and vedolizumab serum trough concentration during vedolizumab SC therapy, will be collected. For evaluation of disease remission at baseline and at control visit, Harvey-Bradshaw index (HBI) for Crohn's disease and Partial Mayo score (PMS) for ulcerative colitis (HBI <5 or PMS <2); or value of fecal calprotectin (<150 µ/g); or Simple Endoscopic Score for Crohn's disease (SES-CD) and Mayo endoscopic subscore (MES) for ulcerative colitis (SES-CD <3 or MES <2), will be used.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older
2. Diagnosis of IBD (UC or CD)
3. Signed informed consent
4. Switched to or planning to switch from vedolizumab IV to vedolizumab SC
5. Disease remission at the time of switch (according to clinical, laboratory or endoscopic parameters)

Exclusion Criteria:

1. Corticosteroid therapy at time of switch from vedolizumab IV to vedolizumab SC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with UC or CD receiving vedolizumab treatment in accordance with the approved SmPC.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Mean Serum Vedolizumab Through Concentration After Switching from Vedolizumab IV to Vedolizumab SC | Up to 12 months from switch
Percentage of Participants in Remission After Switching to Vedolizumab SC | Up to 12 months from switch
  Remission status will be defined by clinical scores (Harvey-Bradshaw index <5 or Partial Mayo score <2), by fecal calprotectin (< 150 mcg/g; if done) or by endoscopic score (SES-CD<3 or Mayo endoscopic subscore<2; if done).
Rate of Hospitalizations After Switching to Vedolizumab SC | Up to 12 months from switch
  Hospitalizations due to inflammatory bowel disease activity or complications will be taken into account.
Rate of Surgery After Switching to Vedolizumab SC | Up to 12 months from switch
  Surgery due to inflammatory bowel disease activity or complications will be taken into account.
Rate of Treatment Change After Switching to Vedolizumab SC | Up to 12 months from switch
  Treatment change is defined as start of corticosteroid therapy, switch to vedolizumab IV again or switch to another biologic or small molecule.

CONTACTS AND LOCATIONS:
Overall Officials: Vlasta Oršić Frič, MD, Principal Investigator — University Hospital Center Osijek
Locations (1):
- Klinički bolnički centar Osijek (University Hospital Center Osijek), Osijek, Croatia